CLINICAL TRIAL: NCT05922267
Title: Comparative Effects of Active Cycle of Breathing Techniques and Slow Expiration With Open Glottis in Lateral Posture in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Comparative Effects of ACBT and Slow Expiration in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0321
Record Dates: First submitted 2023-06-06; First posted 2023-06-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD(chronic obstructive pulmonary disease),; ACBT(active cycle of breathing techniques); ELTGOL
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cycle of breathing technique (Experimental): Try to keep your chest
  * Take a long, slow and deep breath in, through your nose if you can.
  * At the end of the breath in, hold the air in your lungs for 2-3 seconds before breathing
  * Breathe out gently and relaxed, like a sigh. Don't force the air out.
  * Repeat 3 - 5 times.
  * If the patient feels light-headed then it is important that they revert back to the breathing control phase of the cycle
  * Huffing
  Interventions: Other: ACTIVE CYCLE OF BREATHING TECHNIQUES
- SLOW EXPIRATION WITH OPEN GLOTTIS IN LATERAL POSITION (Experimental): The participants in group B will be given slow expiration with open glottis in lateral posture and conventional chest physiotherapy .In this technique, a patient adopts a lateral posture or a lateral decubitus posture. The affected lung is in the dependent position. A patient commences breathing normally, at tidal volumes. They are then instructed to perform a series of slow expirations with an open glottis. Expiration from functional residual capacity to the end of the expiratory reserve volume are encouraged to achieve maximum inflation . To assist in maintaining an open glottis, a mouthpiece may be used, to decrease the degree of airway compression A series of three ELTGOL may be performed, with each series composed of approximately 10 slow and deep expirations. In between each series of maneuvers, a rest period (around 1-2 minutes) is provided, with the patient staying in the same position. A typical treatment lasts for around 20 minutes
  Interventions: Other: SLOW EXPIRATION WITH OPEN GLOTTIS IN LATERAL POSITION

INTERVENTIONS:
Other: ACTIVE CYCLE OF BREATHING TECHNIQUES — The participants in group A will be given ACBT with conventional chest physiotherapy .
  Instruction for patient
  * Try to keep your chest
  * Take a long, slow and deep breath in, through your nose if you can.
  * At the end of the breath in, hold the air in your lungs for 2-3 seconds before breathing
  * Breathe out gently and relaxed, like a sigh. Don't force the air out.
  * Repeat 3 - 5 times.
  * If the patient feels light-headed then it is important that they revert back to the breathing control phase of the cycle
  * Huffing
  Arms: Active cycle of breathing technique
Other: SLOW EXPIRATION WITH OPEN GLOTTIS IN LATERAL POSITION — The participants in group B will be given slow expiration with open glottis in lateral posture and conventional chest physiotherapy .In this technique, a patient adopts a lateral posture or a lateral decubitus posture. The affected lung is in the dependent position. A patient commences breathing normally, at tidal volumes. They are then instructed to perform a series of slow expirations with an open glottis. Expiration from functional residual capacity to the end of the expiratory reserve volume are encouraged to achieve maximum inflation . To assist in maintaining an open glottis, a mouthpiece may be used, to decrease the degree of airway compression A series of three ELTGOL may be performed, with each series composed of approximately 10 slow and deep expirations. In between each series of maneuvers, a rest period (around 1-2 minutes) is provided, with the patient staying in the same position. A typical treatment lasts for around 20 minutes
  Arms: SLOW EXPIRATION WITH OPEN GLOTTIS IN LATERAL POSITION

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by nonreversible airway obstruction. A diagnosis of COPD is determined by clinical assessment of airflow limitation and symptoms such as cough and wheeze; however, the detrimental effect of COPD symptoms on a patient's quality of life is often underestimated. Rehabilitation exercise can lessen the possibility of the progressive exacerbation of the patient's condition, exerting an active role in improving their lung function and the quality of the patients' life .Therefore, Active cycle breathing techniques (ACBT) is a cycle of techniques consisting of breathing control, lower thoracic expansion exercises and the forced expiration technique modifiable for every patient to reduce condition . The effect of ELTGOL on mucus clearance of right and left lungs, especially of peripheral lung areas, in stable patients with COPD . A couple of relaxed breaths and when you are ready go on to your huff. Repeat the huff two or three times until you have the urge to cough. Once you have cleared your chest have a few normal relaxed breaths and start the cycle over again with deep breaths and huffs.

A Randomized clinical trial, subjects with age group between 4O-70 years. In Group -A subjects (n=15) were treated with Active Cycle of Breathing Technique where Group-B subjects (n=15) received ELTGOL training . This study is to compare the effectiveness of ACBT and ELTGOL on improving the Quality Of Life and increasing Functional Capacity in subjects with COPD . Assessment will be done before and after intervention and result will be analyzed using statistical package for social sciences SPSS 20.

ELIGIBILITY:
Inclusion Criteria:

* Both genders (Male and Female)
* 40-70 years
* Diagnosed COPD according to GOLD classification
* Hemodynamically stable patient

Exclusion Criteria:

* Patient with other disorders like cardiac and respiratory disorders
* Carcinoma
* Lung surgery
* Neurological disorders

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Dyspnea scale to assess change in pre and post | base line and fourth week
  Medical Research Council (MRC) chronic dyspnea scale, used for the estimation of disability due to dyspnea, may serve as a simple index of disease severity and extent in patients with lung disease. This scale consists of six questions about perceived breathlessness: category 0, no dyspnea; category 1, slight degree of dyspnea (troubled by shortness of breath when hurrying on the level or walking up a slight hill); category 2, moderate degree of dyspnea (walks slower than people of the same age on the level because of breathlessness); category 3, moderately severe degree of dyspnea (has to stop because of breathlessness when walking at own pace on the level); category 4, severe degree of dyspnea (stops for breath after walking about 100 yards or after a few minutes on the level); category 5, very severe degree of dyspnea (too breathless to leave the house or breathless when dressing or undressing
Peak Flow Meter to assess change in pre and post | baseline and fourth week
  Peak flow meter is mini spirometer which measures the PEFR .The Peak Expiratory Flow Rate (PEFR) is the maximum or peak flow rate that is attained during a forceful expiratory effort after taking a deep inspiration .Its normal range is 250 to 400 . The Peak Expiratory Flow Rate (PEFR) is the maximum or peak flow rate that is attained during a forceful expiratory effort after taking a deep inspiration
BCSS to assess change | baseline and fourth week
  In order to give a rapid and simple means of assessing the severity of respiratory symptoms frequent in COPD patients, the Breathlessness, Cough, and Sputum Scale (BCSS) was created. The BCSS is based on a three-item questionnaire that evaluates the patient's sputum production, coughing, and breathlessness
Oximeter to assess change | baseline and fourth week
  A pulse oximeter measures the amount of oxygen that is carried by your blood. Typically, a little clip is attached to the tip of your finger. (On sometimes, the toe or earlobe are used.) A light beam is projected through the skin using the gadget. By measuring the proportion of your blood that is carrying oxygen, it calculates your oxygen level. Your oxygen saturation, often known as SpO2, is displayed on the screen

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papaporfyriou A, Bakakos P, Hillas G, Papaioannou AI, Loukides S. Blood eosinophils in COPD: friend or foe? Expert Rev Respir Med. 2022 Jan;16(1):35-41. doi: 10.1080/17476348.2021.2011219. Epub 2021 Dec 3. PMID 34821191
- [Background] Fei F, Koffman J, Zhang X, Gao W. Chronic Obstructive Pulmonary Disease Symptom Cluster Composition, Associated Factors, and Methodologies: A Systematic Review. West J Nurs Res. 2022 Apr;44(4):395-415. doi: 10.1177/0193945921995773. Epub 2021 Mar 6. PMID 33682534
- [Background] Zisi D, Chryssanthopoulos C, Nanas S, Philippou A. The effectiveness of the active cycle of breathing technique in patients with chronic respiratory diseases: A systematic review. Heart Lung. 2022 May-Jun;53:89-98. doi: 10.1016/j.hrtlng.2022.02.006. Epub 2022 Feb 27. PMID 35235877
- [Background] Munoz G, de Gracia J, Buxo M, Alvarez A, Vendrell M. Long-term benefits of airway clearance in bronchiectasis: a randomised placebo-controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701926. doi: 10.1183/13993003.01926-2017. Print 2018 Jan. PMID 29326318